CLINICAL TRIAL: NCT05378373
Title: Sustainable Habits for Encouraging Even Teen Sleep (SHEETS): A Digital Intervention to Enhance Sleep and Psychiatric Health in Adolescents
Brief Title: Sustainable Habits for Encouraging Even Teen Sleep
Acronym: SHEETS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00109013; 1R34MH128440-01 (NIH)
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-07

CONDITIONS: Sleep; Psychiatric Health
Keywords: Adolescents; Sleep; Psychiatric Health; Digital Intervention

STUDY DESIGN:
Intervention Model Description: Digital Behavioral Intervention
Who Masked: Participant
Masking Description: Participants will be randomly assigned to one of two interventions, and will not be told which intervention they are assigned to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHEETS Arm 1 (Active Comparator): Participants will receive sleep education-related content on factors that impact sleep, like getting enough exercise.
  Interventions: Behavioral: Garmin, Pattern Health App
- SHEETS Arm 2 (Experimental): Participants will receive sleep education-related content to support good sleep, like setting schedules.
  Interventions: Behavioral: Garmin, Pattern Health App

INTERVENTIONS:
Behavioral: Garmin, Pattern Health App — Wearable sensors will deliver individualized feedback to participants according to their assigned intervention

SUMMARY:
This study will examine the feasibility, acceptability, and effectiveness of two digital sleep interventions in improving sleep regularity and psychiatric health during a critical period of adolescence.

DETAILED DESCRIPTION:
This study will be testing two digital sleep health interventions for adolescents. Adolescents in both conditions will receive sleep education-related content. This project also uses an innovative digital platform and wearable sensors to deliver feedback.

The purpose of this research study is to evaluate a 6-week digital sleep intervention to promote healthy sleep patterns. The study will be broken up into two phases: Phase 1: Focus group participation. Participants and their guardian will be asked to participate in a focus group to get their thoughts/opinions on the intervention. Phase 2: Participants and their guardian will be asked to come to 4 different study visits: baseline, post-intervention, 3 month and 6 month follow up. Participants will be asked to complete questionnaires about demographics, psychiatric health, and sleep patterns. The participants will be asked to wear an ActiGraph watch for 24hrs/day for a week for 4 separate weeks, a Garmin for the duration of the 6-week intervention and keep a sleep diary through an online program.

ELIGIBILITY:
Inclusion Criteria:

* ages 12-14 years
* parent concern on the routines/consistency subscale of the Pediatric Sleep Practices Questionnaire, indicating poor sleep practices (score of 2) in at least one of the following: bedtime consistency, wake time consistency, and bedtime routines;
* ability to speak, read and write in English
* access to internet and smartphone device with capacity to download intervention App (iOS and Android)
* valid email address
* ability to follow written and verbal instructions
* ability and willingness to comply with study procedures.

Exclusion Criteria:

* diagnosed sleep disorder
* psychiatric disorder under treatment (medication and/or therapy) or intellectual disability
* chronic pain condition interfering with sleep
* substance use disorder
* use of medication for sleep (prescription or over-the-counter)
* has a sibling also enrolled/participating in the same study

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Sleep Regularity Index (SRI) | baseline, 6 weeks, 3 months, 6 months
  A measure of sleep regularity collected continuously over 7 days via Actigraphy. The SRI is calculated as the proportion of pairs of time points 24 hours apart that have matching sleep/wake status
Feasibility as measured by Recruitment rate | 6 months
  The number of participants consenting (and assenting) divided by the number who were invited.
Feasibility as measured by Retention Rate | 6 months
  The number of participants who return for each sleep regularity assessment divided by the number who were eligible upon completion of the baseline assessment.
Acceptability as measured by activity completion | 6 months
  The number of participants who complete all weekly sessions divided by the total number of weekly sessions.

SECONDARY OUTCOMES:
Change in Self-Reported Sleep Health | baseline, 6 weeks, 3 months, 6 months
  Self-reported sleep will be assessed via the PROMIS pediatric sleep survey, a 5-point Likert scale ranging from Never to Always. Lower scores indicate better outcomes.
Change in Adolescent Reported Psychiatric Health | baseline, 6 weeks, 3 months, 6 months
  As measured by the Youth Self Report, a 112-item questionnaire, with a 3-point Likert scale ranging from Not True to Very True. Lower scores indicate better outcomes.
Change in Parent Reported Psychiatric Health | baseline, 6 weeks, 3 months, 6 months
  As measured by the Child Behavior Checklist, a 112-item questionnaire, with a 3-point Likert scale ranging from Not True to Very True. Lower scores indicate better outcomes.
Sleep Regularity Index (SRI) as measured by Garmin | 6 weeks
  A measure of sleep regularity collected continuously over 6 weeks via Garmin. The SRI is calculated as the proportion of pairs of time points 24 hours apart that have matching sleep/wake status

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Lunsford-Avery, Ph.D., Principal Investigator — Duke University; Naomi Duke, M.D., Principal Investigator — Duke University
Locations (1):
- Duke Children's Primary Care North Durham, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial (including data dictionaries) will be available for this study after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Data will be accessible by researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Proposals and questions for data access should be directed to NDAHelp@mail.nih.gov. To gain access, data requestors will need to sign a data access agreement at https://nda.nih.gov/nda/access-data-info.html.
URL: https://nda.nih.gov/

DOCUMENTS (1):
  • Informed Consent Form (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT05378373/ICF_000.pdf